CLINICAL TRIAL: NCT00556413
Title: Phase II Study Evaluating the Efficacy and Safety of cétuximab Associated With the Protocol FOLFIRINOX (LV5FU Simplified Combined With Irinotecan and Oxaliplatin) in the First Line Treatment in Patients With Metastatic Colorectal Cancer Expressing EGFR or Not
Brief Title: Cetuximab and Combination Chemotherapy as First-Line Therapy in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000574149; CLCC-ERBIRINOX; INCA-RECF0288; EUDRACT-2005-004746-13; MERCK-CLCC-ERBIRINOX
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ERBIRINOX (Experimental): 5FU + Irinotecan + Oxaliplatine + Cetuximab
  Interventions: Biological: cetuximab; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Biological: cetuximab
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cetuximab together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with combination chemotherapy works as first-line therapy in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response rate in patients with metastatic colorectal cancer treated with cetuximab and FOLFIRINOX chemotherapy comprising oxaliplatin, irinotecan hydrochloride, leucovorin calcium, and fluorouracil as first-line therapy.

Secondary

* Determine the objective response rate in patients treated with this regimen.
* Assess the tolerability of this regimen in these patients.
* Determine the time to response and time to progression in patients treated with this regimen.
* Determine the survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 1-2 hours on days 1 and 8. Patients also receive FOLFIRINOX chemotherapy comprising oxaliplatin IV over 2 hours, irinotecan hydrochloride IV over 30-90 minutes, and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 15 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Metastatic, unresectable disease
* May or may not express the EGFR gene
* Measurable disease, defined as ≥ 1 measurable lesion by MRI or CT scan

  * Lesion must be outside an irradiated area

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy > 3 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Transaminases ≤ 2.5 times ULN (5 times ULN if hepatic metastases are present)
* Creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No peripheral or symptomatic neuropathy ≥ grade 2 (NCI-CTCAE)
* No complete or partial intestinal blockage
* No intestinal inflammatory disease (e.g., Crohn's disease or ulcerative colitis)
* No chronic diarrhea
* No severe unstable cardiac disease (despite treatment)
* No myocardial infarction within the past 6 months
* No neurological or psychiatric illness, including epilepsy or dementia
* No uncontrolled active infection
* No other prior or concurrent malignancy within the past 5 years except for curatively treated basal cell skin cancer
* No psychological, familial, social, or geographic reason that would preclude study follow-up

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic disease

  * Prior fluorouracil-based adjuvant chemotherapy allowed provided it was administered ≥ 4 weeks ago
* At least 4 weeks since prior and no other concurrent experimental therapy
* No prior irinotecan hydrochloride, oxaliplatin, or monoclonal antibody
* No prior intestinal resection (e.g., hemicolectomy or extended resection of the small intestine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-09; Primary Completion 2011-05 (Actual); Study Completion 2011-11-17 (Actual)

PRIMARY OUTCOMES:
Complete response rate | 6 months

SECONDARY OUTCOMES:
Objective response rate | 6 months
Adverse events by using NCI-CTC | 6 months
Time to response | 6 months
Time to progression | 6 months
Survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ychou, MD, PhD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

REFERENCES:
- [Result] Assenat E, Desseigne F, Thezenas S, Viret F, Mineur L, Kramar A, Samalin E, Portales F, Bibeau F, Crapez-Lopez E, Bleuse JP, Ychou M. Cetuximab plus FOLFIRINOX (ERBIRINOX) as first-line treatment for unresectable metastatic colorectal cancer: a phase II trial. Oncologist. 2011;16(11):1557-64. doi: 10.1634/theoncologist.2011-0141. Epub 2011 Oct 20. PMID 22016477